CLINICAL TRIAL: NCT07301606
Title: Static Versus Dynamic Wrist-Hand Splints to Reduce Wrist Spasticity in Subacute Hemiplegic Stroke Patients: A Randomized Control Trial
Brief Title: Static Versus Dynamic Splints for Wrist Spasticity in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Asma Ameer, Physiotherapist, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0030
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Spasticity; Hemiplegia; Post Stroke Recovery
MeSH Terms: conditions — Stroke; Muscle Spasticity; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm 1 (Static wrist-hand splint) (Experimental): Participants in this arm will receive a static wrist-hand splint, which is designed to hold the wrist and fingers in a fixed position. The splint is worn according to the rehabilitation protocol, typically for several hours per day, to help maintain joint alignment, prevent contractures, and reduce wrist flexor spasticity. Participants will undergo wrist spasticity assessments at baseline and at the end of the intervention period.
  Interventions: Device: Static Wrist-Hand Splint
- Arm 2 (Dynamic wrist-hand splint) (Experimental): Participants in this arm will receive a dynamic wrist-hand splint, which applies gentle, graded extension forces to the wrist and fingers while allowing limited movement. The splint is worn according to the rehabilitation protocol, typically for several hours per day, to reduce wrist flexor spasticity and improve wrist positioning. Participants will undergo wrist spasticity assessments at baseline and at the end of the intervention period.
  Interventions: Device: Dynamic Wrist-Hand Splint

INTERVENTIONS:
Device: Static Wrist-Hand Splint — Intervention 1: The static wrist-hand splint is a rigid device that holds the wrist and fingers in a fixed position. It is custom-fitted to each participant and worn according to a defined rehabilitation protocol, typically for several hours per day. The static splint provides continuous support to prevent wrist flexor contractures and reduce spasticity. The primary focus is on maintaining proper joint alignment and minimizing muscle hypertonicity.
  Arms: Arm 1 (Static wrist-hand splint)
Device: Dynamic Wrist-Hand Splint — Intervention 2: The dynamic wrist-hand splint is a device designed to allow controlled, graded wrist and finger extension while limiting excessive flexion. It is custom-fitted to each participant and worn according to a rehabilitation protocol, typically for several hours per day. It permits movement within a safe range while applying gentle extension forces to reduce wrist flexor spasticity. This intervention aims to actively modulate muscle tone while maintaining functional mobility.
  Arms: Arm 2 (Dynamic wrist-hand splint)

SUMMARY:
The goal of this clinical trial is to evaluate whether different types of wrist-hand splints can reduce wrist flexor spasticity in subacute hemiplegic stroke patients. The main questions it aims to answer are:

* Does a dynamic wrist-hand splint reduce wrist spasticity more effectively than a static splint?
* Does one type of splint lead to better functional outcome during use? Researchers will compare participants who receive a static splint with those who receive a dynamic splint to see which splint provides greater improvement in wrist spasticity.

Participants will:

* Wear either a static or dynamic wrist-hand splint according to the assigned study group.
* Undergo wrist spasticity assessments before and after the intervention using a standardized clinical scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years
* Diagnosis of subacute stroke (e.g., 1-6 months post-stroke)
* Presence of wrist flexor spasticity
* Ability to follow simple instructions

Exclusion Criteria:

* Fixed wrist contracture
* Severe pain limiting splint use
* Other neurological or musculoskeletal disorders affecting the upper limb

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Wrist Flexor Spasticity | Baseline to post-intervention (4 weeks)
  Wrist flexor spasticity will be assessed using the Modified Ashworth Scale (MAS). Assessments will be performed at baseline before the intervention and after completion of the intervention period. The primary outcome is the change in MAS score, comparing participants using static versus dynamic wrist-hand splints.

CONTACTS AND LOCATIONS:
Locations (1):
- Markaz Bahali-e- Mazooran, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small number of patients with subacute stroke, and sharing de-identified data could risk participant privacy. Additionally, the data were collected for this specific study and yet no plans have been made to create a broader data repository.

DOCUMENTS (1):
  • Study Protocol (2025-06-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT07301606/Prot_000.pdf